CLINICAL TRIAL: NCT03290495
Title: Electroencephalographic Effects of Ketamine During Isoflurane Maintenance and Recovery
Brief Title: Ketamine Effect on Isoflurane Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hassan, Mamdouh Hassan Mohamed, lecturer of anesthesia and intensive care, Minia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: isoflurane ketamine gamma
Record Dates: First submitted 2017-09-08; First posted 2017-09-25 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Post-anesthesia Recovery
Keywords: ketamine; isoflurane; electroencephalography; maintenance; recovery; anesthesia
MeSH Terms: interventions — Ketamine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Intervention Model Description: An intravenous catheter was placed and normal saline (0.9%) will be infused. Spinal anesthesia will be given. The stability of spinal anesthesia will be assured before propofol injection and at the end of procedure.
  Propofol will be given to facilitate isoflurane inhalation which will be varied between 0.8-1.2percent to keep (BIS) in the range 40-60. Anesthesia will be kept as so for 30 minutes. Then the test drug (either ketamine or saline) will be given slowly, to pressor response in case of ketamine. Anesthesia will be maintained for another 30 minutes then isoflurane is discontinued. Recovery from anesthesia will then be tested.. No other drugs will be routinely given. Development of complications or signs of inadequate anesthesia will cause drop of the case from study and any measures will be taken to insure patient safety and comfort.The patient will be let to recover from anesthesia then transferred to postoperative care unit.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The patients well be randomized to one of the two groups by closed envelope technique. After opening the envelope, the study drug (ketamine 100µg/kg total body weight (Isoket group)) or normal saline ((Isonly) or control group) will be prepared, made up to 10 ml and administered by an assistant in the proper timing. The patient identification will be written on a slip and put back into an envelope and sealed. The person doing the procedure and monitoring along with the patient will be blinded to the dose and nature of solution. The equal volume test solution will be given intravenously by an assistant who was not involved in the administration of anesthesia and monitoring
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- isonly (Active Comparator): This arm will receive spinal anesthesia. then this arm will receive saline during isoflurane anesthesia. this arm will serve as a control group.
  Interventions: Drug: saline
- isoket (Active Comparator): this arm will receive spinal anesthesia. then will receive isoflurane inhalation. during isoflurane inhalation, this arm will receive single injection of ketamine. at end of anesthesia, effect of ketamine on recovery will be monitored.
  Interventions: Drug: ketamine

INTERVENTIONS:
Drug: ketamine — ketamine hydrochloride 250microgram/ ml for iv injection after 30 minutes of stable isoflurane anesthesia
  Other Names: Calypsol
  Arms: isoket
Drug: saline — a similar volume of normal saline 0.9% for intravenous injection instead of ketamine will be given to the control group. this because the attending anesthesiologist will be blinded to the study drugs and aim according to the study proposal.
  Other Names: normal saline, Atsuka
  Arms: isonly

SUMMARY:
Ketamine effect on isoflurane anesthesia This study is designed to study the effect of ketamine on isoflurane anesthesia. As both drugs are hypnotic and are used to cause sleep during surgery and other painful procedures, it was long believed that the actions of two drugs add to each other. For example if a man received both drugs, this man will become awake from anesthesia much later than if this man was given either of them alone.

However recent studies showed that this is not the case and ketamine can cause fast recovery from hypnotic effects of isoflurane. This was confirmed in animals.

The aim of current study is to investigate if this effect applies for humans, using a state of art brain monitoring device in wide use nowadays called BIS or bispectral index. This device can also shed some light on how ketamine can cause, if any, fast recovery from isoflurane anesthesia. Simply, by studying electrical wave coming from brain to head skin.

DETAILED DESCRIPTION:
In an animal study, the authors found that intraperitoneal injection of a sub-anesthetic dose of ketamine amidst isoflurane anesthesia in rats induced early recovery. A finding the authors explained, to be due to increased NMDA mediated increase of acetyl choline secretion in the prefrontal area of rats' brains. This rise, in the authors opinion, antagonized the GABA mediated isoflurane anesthesia resulting in hastened recovery. Meanwhile, the authors found association between hastened recovery and increased Electroencephalographic gamma (EEG γ) wave fronto-parietal projection. This is compatible with cognitive unbinding explanation of unconsciousness during anesthesia.

In current proposed study, the investigator will examine tow hypothesis:

Recovery time:

If the recovery hastening effect of sub anesthetic ketamine on recovery from isoflurane anesthesia is also present in human patients. The assumption will be that ketamine either prolong or has no effect on recovery time from isoflurane anesthesia. The claim well be that ketamine will decrease the recovery time.

Put in statistical terms:

H0: recovery with ketamine ≥ recovery without ketamine. H1: recovery with ketamine ˂ recovery without ketamine. 2. EEG (γ) wave activity: As the investigator will record EEG activity during the procedure via Bispectral monitor, the investigator will analyze the records for presence of enhanced (γ) activity during recovery. the investigator aim is also to detect any significant difference in (γ) wave amplitude or other characteristics between isoflurane only and ketamine group.

The assumption will be that (γ) activity will either show no difference between the two groups or be lower than in ketamine group than isoflurane group during recovery. The claim will be increased (γ) activity with ketamine group during recovery.

Put in statistical terms:

H0: (γ) activity with ketamine ≤ isoflurane only. H1: (γ) activity with ketamine > isoflurane only. N.P: as the sampling frequency of EEG data exported from BIS Vista is 128Hz, the upper limit of the current study of (γ) activity will necessarily be 64Hz.

Sample size calculation:

the mean measured variable of the current study will be the recovery time. Recovery time will be defined as the time between stop of isoflurane inhalation until recovery of verbal response to name called every 30 seconds. A 30% reduction in recovery time in ketamine group as compared with isoflurane is considered to be statically significant enough to reject the null hypothesis of recovery time. According to one study , recovery time from isoflurane only anesthesia is around 12 minutes so the sample size calculation will be as following:

Equation:

n>((ᶻ "1- α ̸2" +ᶻ"1-β" )"2" σ"2" )/δ"2" Where n = sample size required for each group, ᶻ "1-α" = the value for the standard normal distribution for (1-α̸2) percentile, ᶻ "1-β" =the standard normal distribution for 100(1-β) percentile, δ"2" = the difference to detect, σ"2" = the variance in the underling 2 population.

ELIGIBILITY:
Inclusion Criteria:

* Consent: patient must be legally fit to consent. Informed consent will be get from each patient.
* ASA status: I or II.
* Fully conscious at time of induction of anesthesia.
* No history of side effects related to any drugs used in the study.
* Planned surgery can be performed under spinal anesthesia

Exclusion Criteria:

* Incompetence: failure to give informed consent or refusal.
* Neurological or psychiatric disorders
* Addiction
* Recent intake of drugs affecting central nervous system
* ASA state more than II
* Morbid obesity
* Surgery cannot solely performed under spinal anesthesia
* Contraindication to spinal anesthesia as coagulopathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-25 (Actual)

PRIMARY OUTCOMES:
recovery time | Time Frame: 1 hour
  recovery time in this study is defined as time between stop of isoflurane inhalation and recovery of consciousness . this will be assessed by calling the patient first name loudly until the patient verbally respond.time will be recorded in seconds.

SECONDARY OUTCOMES:
gamma wave activity | Time Frame: 2 hour
  EEG will recorded after test drug administration and during recovery. recorded data will be offline analysed for EEG wave activity. the results will be compared between the two study groups.
processed EEG parameters | Time Frame: 2 hour
  this include but not limited to BIS value, spectral edge frequency 95. these value will be online received from BIS monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Mamdouh H Hassan, MD, Principal Investigator — Minia faculty of Medicine. Minia university. Egypt
Locations (1):
- Minia University Hospital (main hospital)-kornish elnil st., Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li D, Hambrecht-Wiedbusch VS, Mashour GA. Accelerated Recovery of Consciousness after General Anesthesia Is Associated with Increased Functional Brain Connectivity in the High-Gamma Bandwidth. Front Syst Neurosci. 2017 Mar 24;11:16. doi: 10.3389/fnsys.2017.00016. eCollection 2017. PMID 28392760
- [Background] Mashour GA. Cognitive unbinding: a neuroscientific paradigm of general anesthesia and related states of unconsciousness. Neurosci Biobehav Rev. 2013 Dec;37(10 Pt 2):2751-9. doi: 10.1016/j.neubiorev.2013.09.009. Epub 2013 Sep 26. PMID 24076246
- [Background] Philip BK, Kallar SK, Bogetz MS, Scheller MS, Wetchler BV. A multicenter comparison of maintenance and recovery with sevoflurane or isoflurane for adult ambulatory anesthesia. The Sevoflurane Multicenter Ambulatory Group. Anesth Analg. 1996 Aug;83(2):314-9. doi: 10.1097/00000539-199608000-00019. PMID 8694311
- [Background] Campbell MJ, Julious SA, Altman DG. Estimating sample sizes for binary, ordered categorical, and continuous outcomes in two group comparisons. BMJ. 1995 Oct 28;311(7013):1145-8. doi: 10.1136/bmj.311.7013.1145. PMID 7580713
- [Background] Florey CD. Sample size for beginners. BMJ. 1993 May 1;306(6886):1181-4. doi: 10.1136/bmj.306.6886.1181. PMID 8499826